CLINICAL TRIAL: NCT00119652
Title: Multicentre, Double-blind, Randomised, Parallel Group, Placebo Controlled, Phase 3 Study of the Efficacy & Safety of Quetiapine Fumarate & Paroxetine as Monotherapy in Adult Patients With Bipolar Depression for 8 Weeks & Quetiapine in Continuation (Abbreviated)
Brief Title: Seroquel in Bipolar Depression Versus SSRI
Acronym: EMBOLDEN II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1447C00134
Record Dates: First submitted 2005-07-06; First posted 2005-07-14 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Bipolar Disorder; Bipolar Depression; Depression
Keywords: Bipolar disorder; bipolar depression; depression
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Quetiapine Fumarate; Paroxetine

INTERVENTIONS:
Drug: quetiapine fumarate (Seroquel)
Drug: paroxetine
Behavioral: mood stabilizing activity

SUMMARY:
The purpose of this study is to determine whether quetiapine is effective and safe in the acute treatment of bipolar depression and whether the effect is maintained when treatment is continued.

ELIGIBILITY:
Inclusion Criteria:

* Male and female out-patients aged 18 to 65 years inclusive
* Diagnosis of Bipolar Disorder (Bipolar I or Bipolar II), most recent episode depressed

Exclusion Criteria:

* Current period of depression lasting less than 4 weeks or more than 12 months
* Use of prohibited medication
* Substance or alcohol dependence or abuse
* Current suicide risk or suicide attempt within 6 months
* Breast feeding or pregnancy
* Clinically relevant disease or clinical finding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 676 (Actual)
Dates: Start 2005-05; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Week 8 assessment in the total score on the Montgomery-Asberg Depression Rating Scale (MADRS)

SECONDARY OUTCOMES:
Secondary variables supportive to the primary objective:
MADRS total score response
MADRS total score remission

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Seroquel Medical Science Director, MD, Study Director — AstraZeneca
Locations (55):
- United States (28):
  - Research Site, Phoenix, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, National City, California
  - Research Site, San Clemente, California
  - Research Site, San Diego, California
  - Research Site, Maitland, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Smyrna, Georgia
  - Research Site, Northfield, Illinois
  - Research Site, Oak Brook, Illinois
  - Research Site, New Orleans, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Glen Burnie, Maryland
  - Research Site, St Louis, Missouri
  - Research Site, Clementon, New Jersey
  - Research Site, New York, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Irving, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Bellevue, Washington
  - Research Site, Kirkland, Washington
- Australia (5):
  - Research Site, Brisbane, Queensland
  - Research Site, Everton Park, Queensland
  - Research Site, Southport, Queensland
  - Research Site, Epping, Victoria
  - Research Site, Malvern, Victoria
- Chile (2):
  - Research Site, Providencia Santiago
  - Research Site, Santiago
- Research Site, Bogotá, Colombia
- Research Site, San José, Costa Rica
- Greece (3):
  - Research Site, Athens
  - Research Site, Thessaloniki
  - Research Site, Tripoli
- Mexico (2):
  - Research Site, México
  - Research Site, Yucatán
- Peru (2):
  - Research Site, Lima
  - Research Site, San Borja
- Romania (4):
  - Research Site, Bucharest
  - Research Site, Galati
  - Research Site, Iași
  - Research Site, Măgura
- South Africa (4):
  - Research Site, Benoni
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Pretoria
- Turkey (Türkiye) (3):
  - Research Site, Gaziantep
  - Research Site, Istanbul
  - Research Site, Manisa

REFERENCES:
- [Derived] McElroy SL, Weisler RH, Chang W, Olausson B, Paulsson B, Brecher M, Agambaram V, Merideth C, Nordenhem A, Young AH; EMBOLDEN II (Trial D1447C00134) Investigators. A double-blind, placebo-controlled study of quetiapine and paroxetine as monotherapy in adults with bipolar depression (EMBOLDEN II). J Clin Psychiatry. 2010 Feb;71(2):163-74. doi: 10.4088/JCP.08m04942gre. Epub 2010 Jan 26. PMID 20122366